CLINICAL TRIAL: NCT00250536
Title: Anabolic Steroids and Exercise in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DK56182 (completed)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: End-Stage Renal Disease; Muscle Weakness
MeSH Terms: conditions — Kidney Failure, Chronic; Muscle Weakness | interventions — Nandrolone Decanoate; Resistance Training

INTERVENTIONS:
Drug: nandrolone decanoate
Behavioral: resistance exercise training

SUMMARY:
This is a study to find out whether an exercise program during dialysis or a drug called nandrolone decanoate can increase muscle size and strenght in patients on dialysis.

DETAILED DESCRIPTION:
Dialysis patients have limited physical functioning as measured by self-reported functioning, peak oxygen consumption, physical performance tests, and tests of muscle strength. A recent study highlighted the severity of debility, reporting that more than one third of hemodialysis patients were unable to perform the normal activities of daily living without assistance. In addition, physical functioning has been shown to be a major determinant of patients' assessment of their global quality of life. Taken together, available evidence suggests that impaired physical functioning is widespread among dialysis patients and profoundly affects their lives. Therefore, interventions to improve functioning in this population have the potential to significantly improve quality of life.

Muscle wasting and weakness are particularly attractive targets for intervention because they are related to loss of function and can be objectively measured and targeted for improvement. Small studies support the possible benefits of two strategies to increase muscle size and strength among patients on dialysis. Anabolic steroids were frequently used to ameliorate the anemia associated with end-stage renal disease prior to the introduction of recombinant erythropoietin, and these agents were noted to cause an increase in serum creatinine along with increases in hemoglobin and hematocrit. More recently, nandrolone decanoate has been shown to increase lean body mass and improve physical performance, and resistance exercise training has been shown to increase strength and improve physical performance. Neither of these preliminary results has been confirmed, nor have the relative benefits of these strategies or their potential additive or synergistic effects been examined. Therefore, we designed a study to compare changes in lean body mass, muscle size and strength, physical performance, and self-reported functioning over a12 week period among hemodialysis patients randomly assigned to one of four groups: 1) nandrolone decanoate, a synthetic testosterone derivative, by weekly intramuscular injection (ND); 2) weekly placebo injections (PL); 3) lower extremity resistance exercise training during dialysis sessions three times per week plus weekly placebo injections (EX); and 4) resistance exercise plus nandrolone injections weekly (EX+ND).

ELIGIBILITY:
Inclusion Criteria:

* end-stage renal disease on hemodialysis for 3 or more months

Exclusion Criteria:

* inadequate dialysis; Kt/V <1.2
* nonadherent to dialysis treatments; missing >2 dialysis sessions in the month prior to screening
* catabolic state; HIV with opportunistic infection in the last 3 months, malignancy, or infection requiring intravenous antibiotics within 2 months prior to screening
* unable to give informed consent
* active intravenous drug use
* contraindications to resistance exercise; myocardial infarction within 6 months, active angina, uncompensated congestive heart failure, orthopedic or musculoskeletal limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2000-03; Study Completion 2004-10

PRIMARY OUTCOMES:
Primary outcomes included change in lean body mass measured by dual-energy X-ray absorptiometry, quadriceps muscle cross-sectional area (CSA) measured by MRI, and knee extensor muscle strength.

SECONDARY OUTCOMES:
Secondary outcomes included changes in physical performance, self-reported physical functioning, and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten L Johansen, MD, Principal Investigator — University of California, San Francisco, San Francisco VA Medical Center

REFERENCES:
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639